CLINICAL TRIAL: NCT02907515
Title: Maintenance and Cost Effectiveness of CM-LOC Resin Matrix Versus Ball Nylon Matrix Attachment Retaining Single Implant Mandibular Complete Overdentures
Brief Title: Maintenance and Cost Effectiveness of Cendres Metaux Locator (CM-LOC) Resin Matrix Versus Ball Nylon Matrix Attachment Retaining Single Implant Mandibular Complete Overdentures
Acronym: MCRB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Ahmed Naguib, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CEBD-CU-2016-09-196
Record Dates: First submitted 2016-09-08; First posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Completely Edentulous
Keywords: single implant retained mandibular overdenture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cm-loc attachment (Experimental): cm-loc attachment is a new attachment for dental implants and connect to the denture with resin matrix as housing
  Interventions: Device: cm-loc attachment
- ball attachment (Active Comparator): ball attachment is the most common attachment for dental implants and connect to the denture by nylon cap and metal housing
  Interventions: Device: ball attachment

INTERVENTIONS:
Device: cm-loc attachment — cm-loc is a new implant attachment mechanism with resin matrix housing to retain the overdenture
  Arms: cm-loc attachment
Device: ball attachment — ball attachment is the gold slandered attachment mechanism with nylon cap and metal housing to retain the overdenture
  Arms: ball attachment

SUMMARY:
The single implant overdenture (IOD) represent the simplest form of IODs compared to the 2 IOD which is the traditional gold standard IOD treatment option. Mandibular single-implant overdentures are proven to be a successful treatment option for older edentulous adults but we need to know if the CM-LOC attachment will retain its superiority over the ball attachments intraorally regarding the prosthetic complications in single implant retained overdenture like in 2 IOD

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous male or female patients between the ages of 50 to 69.
* No contraindications for implantation.
* Each patient has to perform both a random blood sugar and Glycosylated Hemoglobin analysis. Patients with a Glycosylated hemoglobin test HbA1c up to 8% and a normal blood sugar level (79 to 110) or controlled diabetic patients (90-130 fasting according to American Association of Diabetes) will be included.
* Sufficient bone width (≥ 6 mm) in the anterior region to place an implant. It could be either normally present or achieved by bone plateauing. This will be confirmed by cone beam computed tomographic (CBCT) scans.
* Residual bone height ranging from 11-20 mm with the lowest vertical height in the midline of the mandible not less than 13 mm (Class II or III according to McGarry et al[1] 1999). This will be confirmed by the CBCT.
* Patients seeking to install a single symphyseal implant and for whom new dentures will be constructed.
* Patients, who are dissatisfied with the retention and stability of their technically satisfactory dentures.
* Patients, who already have existing maxillary and mandibular complete dentures, and after examination of the mandibular dentures, it is found that there are technical problems with regard to denture design and/or occlusion; then new maxillary and mandibular dentures will be fabricated
* All patients should have adapted to their dentures for at least six weeks before being included in the trial.
* Patients providing written informed consents to participate in the trial and this will be done before the scheduled date for implant installation.

Exclusion Criteria:

* Patients with a systemic or local contra-indication for implant placement.
* Satisfied patients with the retention of their mandibular denture as well as unsatisfied patients with their maxillary denture.
* Patient with a mandibular denture height less than 6 mm between the base of the denture and the incisal edge of the central incisors (as measured by a caliper) or with 12 mm crown height space as measured by a ruler from the incisal edge till the crest of the ridge. This will be done from a putty index of the diagnostic set up.
* Incompliant and not cooperative patients.
* Patients smoking more than 10 cigarettes per day

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
number of prosthodontic Maintenance events | 1 year
  the number of the patient visits to the doctor to make maintenance for his implant supported overdenture

SECONDARY OUTCOMES:
cost effectiveness (which treatment will cost less money) | 1 year
  amount of usa dollars scale spent on either attachment cm-loc or ball attachment in fabrication and maintenance

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo Universty, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No